CLINICAL TRIAL: NCT06053996
Title: Hepatopulmonary Radio-sterilization Combined With Checkpoint Inhibition, a Proof-of-concept Phase II Clinical Trial in Colorectal Cancer
Brief Title: Hepatopulmonary Radio-sterilization With Immunotherapy
Acronym: TROS-8
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-23-0497-OM-CTIL
Record Dates: First submitted 2023-08-07; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Colon Cancer; Liver Metastasis Colon Cancer; Rectal Cancer
Keywords: radiation; radiotherapy; SBRT; immunotherapy; Stereotactic ablative radiotherapy (SABR)
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: radiation to hepatic and pulmonary metastases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MSI-H mCRC (Experimental): high dose radiation therapy (SBRT) targeted to the lung and liver metastases
  Interventions: Radiation: Hepatopulmonary radio-sterilization
- MSS mCRC. (Experimental): high dose radiation therapy (SBRT) targeted to the lung and liver metastases
  Interventions: Radiation: Hepatopulmonary radio-sterilization

INTERVENTIONS:
Radiation: Hepatopulmonary radio-sterilization — Hepatopulmonary radio-sterilization - ablation of hepatic and pulmonary metastases

SUMMARY:
In this protocol the investigators aim to overcome hepatic-pulmonary metastases-induced resistance to immunotherapy through high dose radiation therapy (SBRT) targeted to the metastases themselves, aiming, when possible, to ablate all macroscopic disease in these organs.

DETAILED DESCRIPTION:
A number of recent reports have noted the relative resistance of liver metastases to immunotherapy across a range of cancer types1,2, including mCRC. In two studies of MSS mCRC using a combination of PD-1 and CTLA-4 inhibitors there was a marked difference in response rate between subjects with and without liver metastases, 0% vs 42% in the study of Bullock et al3, and 0% versus 36% in the study by Fakih et al4. The proposed mechanism is a macrophage-induced T cell death occurring within hepatic metastases, leading to systemic imunosupression5. Furthermore, these investigators demonstrated that in preclinical models of MSS mCRC, liver-metastasis directed radiotherapy eliminates immunosuppressive hepatic macrophages, increases hepatic T cell survival and reduces hepatic siphoning of T cells, thereby abolishing the immunotherapy resistance induced by liver metastasis5. Conversely, liver irradiation in the absence of metastases was ineffective5.

Similarly, in microsatellite instability high mCRC the presence of liver metastases is associated with a poor response to immunotherapy6. In a retrospective analysis of 161 MSI High mCRC patients treated with immunotherapy, pooling data from MD Anderson and Sheba, the presence of liver and lung metastases was associated with a reduced PFS, with a HR of 2.6 and 2.4, respectively (submitted for publication).

In this protocol the investigators aim to overcome hepatic-pulmonary metastases-induced resistance to immunotherapy through high dose radiation therapy (SBRT) targeted to the metastases themselves, aiming, when possible, to ablate all macroscopic disease in these organs.

ELIGIBILITY:
Inclusion Criteria:

Disease factors

* Histologically- or cytologically-confirmed diagnosis of colorectal cancer (CRC).
* Metastatic or recurrent CRC, deemed surgically or medically unresectable.
* Subjects who are candidates to receive immunotherapy, whether MSS or MSI-high.
* Subjects who have liver and / or lung metastases amenable to SBRT.

General considerations

* Age ≥18 years.
* ECOG performance status ≤1 (Karnofsky ≥70%, see Appendix A).
* Life expectancy of ≥ 3 months
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count ≥1,500/mcL
* platelets ≥100,000/mcL
* hemoglobin ≥ 9.0 g/dL
* total bilirubin ≤ 1.5 x ULN except subjects with Gilbert Syndrome must have a total bilirubin level < 3.0 mg/dL).
* AST(SGOT)/ALT(SGPT) ≤2.0 × institutional upper limit of normal
* creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 50 mL/min (using the Cockcroft Gault formula)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of treatment.
* Signed Written Informed Consent
* Subjects must have signed and dated an IRB approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.

Exclusion Criteria:

- Disease factors / Tumor characteristics

• Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.

Previous treatments and trials

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 3 weeks of the first dose of treatment.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Comorbidities, medications and immune modulation agents

* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with type I diabetes mellitus, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects that require intermittent use of bronchodilators or local steroids, e.g., inhaled or topical steroids, at a dose of less than the equivalent of 10mg prednisone daily, would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.
* History of allergy or hypersensitivity to any study drug components, to compounds of similar chemical or biologic composition
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years
  Safety and tolerability

SECONDARY OUTCOMES:
6 month PFS | 6 months
  progression free survival at 6 months
Overall survival (OS) | 4 years
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Margalit, MD PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No